CLINICAL TRIAL: NCT02981186
Title: Comparison of Visual Outcomes After Implantation of the POD AY GF F (PhysIOL) and the POD AY 26P F (PhysIOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1603
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Cataract; Lens Opacity
Keywords: Intraocular Lens; trifocal; cataract; PhysIOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL Implantation experimental (Experimental): Implantation of POD F GF in one of the eyes of the study subject
  Interventions: Device: IOL implantation experimental
- IOL Implantation Comparator (Active Comparator): Implantation of POD F in the contralateral eye of the study subject
  Interventions: Device: IOL implantation comparator

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of trifocal IOL POD F GF consisting of hydrophobic material
  Arms: IOL Implantation experimental
Device: IOL implantation comparator — Implantation of trifocal IOL POD F consisting of hydrophilic material
  Arms: IOL Implantation Comparator

SUMMARY:
The study is a prospective randomised controlled study. The patients get monolateral IOL implantation of POD F GF and POD F in the contralateral eye. Both IOLs are trifocal IOLs consisting of the same optical design. The difference between the IOLs is the material (hydrophilic and hydrophobic).

To decide which eye receives POD F and which eye receives POD F GF, a randomization table will be provided to the principle investigator.

DETAILED DESCRIPTION:
The examinations consist of visual acuity data, contrast sensitivity exams and slitlamp examinations.

Follow up will be up to 6 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous Eyes with no comorbidity
* Patient older than 50 years old
* Regular corneal astigmatism <0.75 dioptres by an automatic keratometer (regularity determined by the topography of the keratometry) or <1.0 dioptres if the steep axis of cylinder is between 90° and 120°
* Spontaneously emitting the desire for spectacle independence after surgery and with realistic expectation.
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Unrealistic expectation
* Irregular astigmatism
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Visual Acuity at far, near and intermediate distance | 6 months postoperative
  ability to read letters at different distances

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Nagy, MD, Principal Investigator — Semmelweis University - Department of Ophthalmology
Locations (1):
- Semmelweis University - Department of Ophthalmology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No